CLINICAL TRIAL: NCT03760601
Title: Intrusive Memories of Trauma Experienced by Young Refugees: Using Single Case Experimental Design to Investigate a Brief Cognitive Intervention Involving Computer Gameplay: An Extension
Brief Title: A Brief Cognitive Intervention After Intrusive Memories of Trauma With Young Refugees: An Extension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Emily Holmes, Professor Emily Holmes, Karolinska Institutet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018/2149-32
Record Dates: First submitted 2018-11-19; First posted 2018-11-30 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Intrusive Memories of Trauma, Symptom of Post Traumatic Stress Disorder (Criterion B1)

STUDY DESIGN:
Intervention Model Description: Single case experimental AB design with optional replication (ABAB)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline phase ('A') (No Intervention): Measurements collected in a pen-and-paper diary four times a day (morning, afternoon, evening and night) over one week for the primary outcome (occurrence of intrusive memories of trauma). Individual baseline phases will be used as control periods.
- Intervention phase ('B') (Experimental): A one-session intervention with a researcher including a simple cognitive task (a memory cue, 10 minutes time gap and ca. 20 minutes of Tetris game-play) followed by instructions to engage in the task selfguided over the subsequent week. Measurements collected in a pen-and-paper diary four times a day over one week following the intervention for the primary outcome (occurrence of intrusive memories of trauma).
  Interventions: Behavioral: Brief cognitive intervention

INTERVENTIONS:
Behavioral: Brief cognitive intervention — A one-session intervention with a researcher including a simple cognitive task (a memory cue, 10 minutes time gap and ca. 20 minutes of Tetris game play) with instructions to engage in the task self-guided in the subsequent week.
  Arms: Intervention phase ('B')

SUMMARY:
This research study is designed to investigate the use of a simple cognitive task (a memory cue and 10 minute time gap, followed by playing the computer game "Tetris") for decreasing the number of intrusive memories of trauma among young refugees and asylum seekers. The design is a single case experimental AB design with optional replication (ABAB). Participants will aim to complete a no-intervention phase ('A': baseline phase) of one week followed by a one-week intervention phase ('B'), including a one-session intervention with a researcher comprising the simple cognitive task, followed by instructions to continue to use the technique self-guided in the subsequent week. Follow ups are conducted after each week to monitor the occurrence of intrusive memories of trauma in a pen-and-paper diary. It is predicted that participants will report fewer intrusive memories during the intervention phase than during the preceding baseline phase.

DETAILED DESCRIPTION:
This research study follows from ClinicalTrials.gov ID: NCT03525158, with a focus on the ABAB design and adding additional questions e.g. on concentration, emotion and functioning, and with the possibility of focusing on 1 intrusive memory at a time with associated distress ratings as part of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Refugee or asylum seeker
* Experiencing intrusive memories of trauma
* Have access to a smartphone
* Able to speak or read the study material in Swedish, English, Arabic or Farsi
* Able to attend five to six meetings with a researcher

Exclusion Criteria:

* Exhibit psychotic symptoms or other symptoms of severe mental illness

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Change in number of intrusive memories of trauma | Change between baseline week 1 and Intervention week 1
  Number of intrusive memories of traumatic event recorded by participants in a diary daily (morning, afternoon, evening and night) over one week.

SECONDARY OUTCOMES:
Feasibility and acceptability ratings for using a smartphone game-play intervention | Intervention week 1
  Feasibility and Acceptability of the intervention assessed with 10 self-rated items, e.g. "Would you recommend playing Tetris to a friend?". Scores range from 0 - 10 with higher scores indicating greater acceptability/ feasibility.
Feasibility and acceptability - open ended questions | Intervention week 1
  Two items with open-ended follow-up questions: "How did you feel about playing Tetris after you had an intrusive memory?" and "Why"? or "How much would you prefer an intervention that is delivered by a computer/ smartphone compared to seeing a doctor/psychologist in person?" and "Why"?
Self-guided intervention adherence - usage of the gameplay intervention in daily life | Intervention week 1
  Usage of the gameplay intervention assessed with 4 self-rated items: 1. Did you play Tetris in the last week since the last meeting? (Yes/No). 2. If yes, how many days did you play Tetris in the last week since we first practiced the game together? 3. How long did you spend playing Tetris at a time? (<10 min - >30 min), 4. How often did you manage to play Tetris after you experienced an intrusive memory? (11-point scale; 0 = not at all; 10 = every time).
Impact of intrusive memories on concentration, control, sleep and stress - ratings | Baseline week 1 and Intervention week 1
  A bespoke measure of 6 self-rated items to assess the impact of intrusive memories on concentration, control, sleep and stress (all rated on an 11-point scale): 2 items assessing experienced concentration difficulties due to intrusive memories and in general ( high scores indicating more concentration difficulties);1 item assessing feeling of control over intrusive memories (0 = no control; 10 = in full control); 2 items assessing sleep disturbances due to intrusive memories (higher scores indicating more sleep disturbance); and 1 item assessing to what degree intrusive memories affected stress levels (0 = not at all; 10 = affected very much).
Rating of how long intrusive memories disrupted concentration on average | Baseline week 1 and Intervention week 1
  1 item assessing for how long intrusive memories disrupted concentration on average (<1 minute - > 60 minutes)
Impact of intrusive memories - open ended questions | Baseline week 1 and Intervention week 1
  Two open-ended questions are included: "How do intrusive memories interfere with your concentration?" and "How do intrusive memories interfere with your ability to settle in to this country and learn new skills, e.g. a new language?"
Impact of the intervention on concentration, emotion and functioning - ratings | Intervention week 1
  A bespoke measure comprising 3 self-rated items to assess the impact of the intervention on concentration, emotion and functioning at the time of playing (11-point scale, 0= not helpful, 10= very helpful).
Subjective impact of the intervention - open ended questions | Intervention week 1
  2 open ended questions about the subjective impact of the intervention in the shorter, and longer term: "How would you describe the impact of this intervention in the short term?"; "How would you describe the impact of this intervention in the longer term"?
World Health Organization Disability Assessment Schedule 2.0 (WHODAS) | Baseline week 1 and intervention week 1
  A 12 item self-rated questionnaire asking about difficulties due to health conditions, including mental or emotional problems. Scores range from 1 to 5 where 1=none and 5=extreme or cannot do.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Holmes, Prof, Principal Investigator — Karolinska Institutet
Locations (1):
- Swedish Language Classes for Refugees, Clinics, Stockholm, Sweden

REFERENCES:
- [Result] Kanstrup M, Kontio E, Geranmayeh A, Olofsdotter Lauri K, Moulds ML, Holmes EA. A single case series using visuospatial task interference to reduce the number of visual intrusive memories of trauma with refugees. Clin Psychol Psychother. 2021 Jan;28(1):109-123. doi: 10.1002/cpp.2489. Epub 2020 Jul 6. PMID 32525244